CLINICAL TRIAL: NCT03899506
Title: Prospective Observational Investigation of Olanzapine Versus Midazolam for the Treatment of Acute Undifferentiated Agitation in the Emergency Department
Brief Title: Olanzapine Versus Midazolam for Agitation
Acronym: OvM
Status: Terminated | Type: Observational
Why Stopped: Investigator Voluntary Pause
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Lauren Klein, Principal Investigator, Hennepin Healthcare Research Institute
Other Study IDs: HSR #18-4521
Record Dates: First submitted 2018-06-28; First posted 2019-04-02 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Agitation,Psychomotor
MeSH Terms: conditions — Psychomotor Agitation | interventions — Olanzapine; Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Olanzapine: Patients receiving 10 mg IM Olanzapine per the ED protocol
  Interventions: Drug: Olanzapine
- Midazolam: Patients receiving 5 mg IM Midazolam per the ED protocol
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Olanzapine — Patients receiving Olanzapine per the ED protocol
  Groups: Olanzapine
Drug: Midazolam — Patients receiving Midazolam per the ED protocol
  Groups: Midazolam

SUMMARY:
The goal of this research investigation is to conduct a prospective observation of the comparative efficacy of midazolam versus olanzapine for the treatment of acute undifferentiated agitation in the emergency department.

DETAILED DESCRIPTION:
The goal of this research investigation is to conduct a prospective observation of the comparative efficacy of midazolam versus olanzapine for the treatment of acute undifferentiated agitation in the emergency department.

In the summer of 2017, the ED implemented a treatment protocol as a quality improvement initiative. The investigators performed observational research on this protocol and identified that haloperidol and ziprasidone were inferior to midazolam and olanzapine for treating agitation in our Department.

The comparison between olanzapine and midazolam, however, was inconclusive. It is possible that this is due to inadequate power, so the question of whether olanzapine or midazolam is superior is still unknown.

Because the department continues to strive to achieve the best care for this patient population, in the Summer of 2018 the ED is going to initiate a second ED treatment protocol of olanzapine and midazolam, based on the results of our 2017 protocol.

All patients requiring chemical sedation for will receive olanzapine as the initial treatment for agitation for 6 weeks, followed by midazolam as the initial treatment for agitation for 6 weeks. These patients will be observed by research staff.

This is a clinical care quality improvement protocol. The clinical protocol is not research. The research component is the observation of this clinical care protocol.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients
* Patients 18 years and older
* Patients with acute undifferentiated agitation requiring chemical sedation at the discretion of the attending emergency physician will be observed.

Patients meeting these criteria who receive medications in the ED will be observed by research staff, evaluating efficacy and safety of the administered medication.

Exclusion Criteria:

- There are no exclusion criteria per se as this is only observational research. The decision to administer the medication is at the discretion of the physician. Research protocols are only such that we are observing the efficacy and safety, which coincides the quality improvement purposes of this clinical protocol. Patients will be provided an Information Sheet and can opt to have their data removed.

Patients who are prisoners, children, will NOT have their data collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ED patients with agitation who receive a medication per protocol at the discretion of ED providers
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients Adequately Sedated at 15 minutes | 15 minutes
  Proportion of patients who achieve an AMSS score of < 1 at 15 minutes

SECONDARY OUTCOMES:
Proportion of Patients Adequately Sedated at 30 minutes | 30 minutes
  Proportion of patients who achieve an AMSS score of < 1 at 30 minutes
Proportion of Patients Adequately Sedated at 60 minutes | 60 minutes
  Proportion of patients who achieve an AMSS score of < 1 at 60 minutes
Proportion of Patients Adequately Sedated at 120 minutes | 120 minutes
  Proportion of patients who achieve an AMSS score of < 1 at 120 minutes
Safety Events | 120 minutes
  Proportion of patients who experience respiratory depression, hypotension, extrapyramidal side effects

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Klein, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No